CLINICAL TRIAL: NCT04701944
Title: Clinical Study of Pregnant Women With COVID-19: A Retrospective Review of Medical Records at Strasbourg University Hospitals
Brief Title: Clinical Study of Pregnant Women With COVID-19
Acronym: PregWom-Covid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7794
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
Keywords: COVID-19; COVID-19 Pandemic; Sars-cov-2; Pregnant women
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A new pandemic, COVID-19, has spread rapidly around the world. She does not spare pregnant women. Little is known about the clinical course of pregnant women infected with COVID-19. As of April 1, 2020, six case series and one case report for a total of 61 pregnancies affected by COVID-19, all from the pandemic epicenter in China, except for one state case report -Unis, have been published. These preliminary reports suggest that pregnant women are not more seriously affected than the general population and show a certain gap with what we have observed in the care of pregnant women at HUS. For these reasons, additional information, especially from parts of the world other than China, as the severity of the disease can vary from country to country, is urgently needed to determine whether pregnant women with the disease of COVID-19 will not present with severe pneumonia to COVID-19.

ELIGIBILITY:
Inclusion criteria:

* Adult woman (≥18 years old)
* Pregnant woman
* Suffering from a confirmed or suspected COVID-19 infection
* Patient who has been medically treated at Strasbourg University Hospitals as well as for his newborn baby, between 03/01/2020 and April 30, 2020
* Woman having given, after information, her agreement for the reuse of her data for the purposes of this research

Exclusion criteria:

* Patient who expressed her opposition to participating in the study
* Patient under guardianship or under guardianship
* Patient under legal protection

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant woman suffering from a confirmed or suspected COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-04-21 (Estimated); Study Completion 2021-04-21 (Estimated)

PRIMARY OUTCOMES:
A retrospective review of the medical records of pregnant women with COVID-19 at the University Hospitals of Strasbourg | Files analysed retrospectively from March 01, 2020 to April 30, 2020 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DERUELLE, MD, PhD, Study Director — Department of Gynecology-Obstetrics and Fertility - Strasbourg University Hospitals
Locations (1):
- Department of Gynecology-Obstetrics and Fertility - Strasbourg University Hospitals, Strasbourg, France